CLINICAL TRIAL: NCT01452347
Title: A Randomised, Phase II Study to Evaluate the sAfety and Pharmacokinetics of oraL dabIGatran Etexilate in Patients After Heart Valve replacemeNt
Brief Title: Dabigatran Etexilate in Patients With Mechanical Heart Valves
Acronym: RE-ALIGN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1160.113; 2010-022685-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-07

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases | interventions — Warfarin; Dabigatran

ARMS (2):
- Dabigatran etexilate (Experimental): Patient dose dependent on screening CrCl levels and TT
  Interventions: Drug: dabigatran etexilate intermediate dose; Drug: dabigatran etexilate low dose; Drug: dabigatran etexilate high dose
- warfarin (Active Comparator): warfarin doses to maintain INR levels
  Interventions: Drug: warfarin 1mg; Drug: warfarin 5mg; Drug: warfarin 3mg

INTERVENTIONS:
Drug: warfarin 1mg — comparator warfarin
  Arms: warfarin
Drug: dabigatran etexilate intermediate dose — active treatment (medium)
  Arms: Dabigatran etexilate
Drug: dabigatran etexilate low dose — active treatment (low)
  Arms: Dabigatran etexilate
Drug: warfarin 5mg — comparator warfarin
  Arms: warfarin
Drug: dabigatran etexilate high dose — active treatment (high)
  Arms: Dabigatran etexilate
Drug: warfarin 3mg — comparator warfarin
  Arms: warfarin

SUMMARY:
To validate the dosing algorithm for dabigatran etexilate in patients receiving a mechanical heart valve.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 18-75
2. Patients who have received a bileaflet mechanical heart valve

Exclusion criteria:

1. Prior valve surgery
2. Uncontrolled hypertension
3. severe renal impairment
4. active liver disease
5. increased risk of bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (40):
- Belgium (5):
  - 1160.113.32003 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.113.32007 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.113.32002 Boehringer Ingelheim Investigational Site, Genk
  - 1160.113.32005 Boehringer Ingelheim Investigational Site, Ghent
  - 1160.113.32001 Boehringer Ingelheim Investigational Site, Leuven
- Canada (7):
  - 1160.113.11002 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.113.11006 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1160.113.11001 Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - 1160.113.11009 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.113.11011 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1160.113.11012 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1160.113.11007 Boehringer Ingelheim Investigational Site, Toronto, Ontario
- Czechia (5):
  - 1160.113.42002 Boehringer Ingelheim Investigational Site, Brno
  - 1160.113.42005 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 1160.113.42003 Boehringer Ingelheim Investigational Site, Olomouc
  - 1160.113.42004 Boehringer Ingelheim Investigational Site, Ostrava
  - 1160.113.42001 Boehringer Ingelheim Investigational Site, Prague
- Denmark (2):
  - 1160.113.45001 Boehringer Ingelheim Investigational Site, Copenhagen
  - 1160.113.45002 Boehringer Ingelheim Investigational Site, Odense C
- France (4):
  - 1160.113.33004 Boehringer Ingelheim Investigational Site, Bron
  - 1160.113.33001 Boehringer Ingelheim Investigational Site, Paris
  - 1160.113.33002 Boehringer Ingelheim Investigational Site, Pessac
  - 1160.113.33003 Boehringer Ingelheim Investigational Site, Rennes
- Germany (6):
  - 1160.113.49001 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.113.49002 Boehringer Ingelheim Investigational Site, Essen
  - 1160.113.49008 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1160.113.49004 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1160.113.49003 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1160.113.49010 Boehringer Ingelheim Investigational Site, Witten
- Netherlands (3):
  - 1160.113.31001 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.113.31002 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.113.31004 Boehringer Ingelheim Investigational Site, Breda
- Norway (2):
  - 1160.113.47002 Boehringer Ingelheim Investigational Site, Bergen
  - 1160.113.47001 Boehringer Ingelheim Investigational Site, Oslo
- Poland (3):
  - 1160.113.48004 Boehringer Ingelheim Investigational Site, Gdansk
  - 1160.113.48003 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.113.48001 Boehringer Ingelheim Investigational Site, Wroclaw
- Sweden (3):
  - 1160.113.46004 Sahlgrenska Universitetssjukhuset, Gothenburg
  - 1160.113.46003 Skånes Universitetssjukhus Lund, Lund
  - 1160.113.46001 Akademiska Sjukhuset, Uppsala

REFERENCES:
- [Derived] Eikelboom JW, Connolly SJ, Brueckmann M, Granger CB, Kappetein AP, Mack MJ, Blatchford J, Devenny K, Friedman J, Guiver K, Harper R, Khder Y, Lobmeyer MT, Maas H, Voigt JU, Simoons ML, Van de Werf F; RE-ALIGN Investigators. Dabigatran versus warfarin in patients with mechanical heart valves. N Engl J Med. 2013 Sep 26;369(13):1206-14. doi: 10.1056/NEJMoa1300615. Epub 2013 Aug 31. PMID 23991661

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 patients were not entered/randomized
Groups:
- Dabigatran Etexilate (DE): Oral administration of 1 capsule of 150 mg (150 mg), 2 capsules of 110 mg (220 mg), or 2 capsules of 150 mg (300 mg) twice daily
- Warfarin: Oral administration of Warfarin 1mg, 3mg and 5 mg according to target international normalised ratio (INR), as recommended in guidelines, and deemed appropriate by investigator
Period: Overall Study
Arm/Group | Dabigatran Etexilate (DE) | Warfarin
Started | 168 | 84
Completed | 151 | 77
Not Completed | 17 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Non compliance protocol | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Not treated | 6 | 3
Not completed — Other reason not defined above | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TRT): The set of patients who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate (DE) | Warfarin | Total
Number analyzed (Participants) | 162 | 81 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.2) | 55.8 (10.2) | 56.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 26 | 86
  Male | 102 | 55 | 157

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Observed and Predicted Trough Dabigatran Plasma Concentrations at Steady State (C Trough,ss) at Week 1
Description: Comparisons between dabigatran trough plasma levels as predicted by simulations to those observed in the study are performed to validate the dosing algorithm for Dabigatran Etexilate (DE) .
  Despite the primary endpoint only being assessed in patients who received dabigatran etexilate, Warfarin was included as a comparator treatment in this study in order to facilitate informal comparisons of outcome events, and to look for efficacy signals in this previously unexplored population.
Time Frame: Week 1
Population: Pharmacokinetic set (PKS):Patients were included in the PKS if they were treated with DE, had at least 1 evaluable C trough,ss value and had a non-missing value for gender, age and Creatinine clearance(CrCl) level. Patients who had any important Protocol Violations that may have affected PK data were excluded from the PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Observed: This includes the observed Ctrough,ss value for all patients in the pharmacokinetic set (PKS) who have a corresponding predicted value.
- Predicted: This includes the predicted Ctrough,ss value for all patients in the PKS who have a corresponding observed value.
Arm/Group | Observed | Predicted
Number analyzed (Participants) | 130 | 130
ng/mL | 73.86 (43.9) | 99.52 (43.9)
Statistical Analysis 1: Comparison: Observed vs Predicted; Null hypothesis: "The difference of the population average responses was either ≤ to the lower bound or ≥ to the upper bound of the acceptance range" . Alternative hypothesis: "The difference of the population average responses was both > than the lower bound and < than the upper bound of the acceptance range" [Note: The acceptance range for the geometric mean is 80-125%]; Test type: Superiority or Other; ANOVA; The Ctrough,ss (predicted or observed) was log transformed (natural logarithm) prior to fitting the ANOVA model; Adjusted Geometric Mean ratio = 74.22, 95% CI [68.08 to 80.91], Standard Error of Mean 1.05 — The standard error of the mean is actually the geometric standard error. (Observed vs Predicted)

2. Primary Outcome: Comparison of Observed and Predicted Trough Dabigatran Plasma Concentrations (C Trough,ss) at Week 2
Description: Comparisons between dabigatran trough plasma levels as predicted by simulations to those observed in the study are performed to validate the dosing algorithm for Dabigatran Etexilate (DE).
  Despite the primary endpoint only being assessed in patients who received dabigatran etexilate, Warfarin was included as a comparator treatment in this study in order to facilitate informal comparisons of outcome events, and to look for efficacy signals in this previously unexplored population.
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Observed: This includes the observed Ctrough,ss value for all patients in the PKS who have a corresponding predicted value.
Arm/Group | Observed | Predicted
Number analyzed (Participants) | 26 | 26
ng/mL | 84.08 (40.2) | 99.55 (40.2)
Statistical Analysis 1: Comparison: Observed vs Predicted; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; The Ctrough,ss (predicted or observed) was log transformed (natural logarithm) prior to fitting the ANOVA model; Adjusted Geometric Mean ratio = 84.46, 95% CI [70.32 to 101.44], Standard Error of Mean 1.11 — The standard error of the mean is actually the geometric standard error. (Observed vs Predicted)

3. Primary Outcome: Comparison of Observed and Predicted Trough Dabigatran Plasma Concentrations (C Trough,ss) at Week 4
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Observed | Predicted
Number analyzed (Participants) | 112 | 112
ng/mL | 104.43 (34.3) | 109.36 (34.3)
Statistical Analysis 1: Comparison: Observed vs Predicted; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; The Ctrough,ss (predicted or observed) was log transformed (natural logarithm) prior to fitting the ANOVA model; Adjusted Geometric Mean ratio = 95.50, 95% CI [88.69 to 102.84], Standard Error of Mean 1.05 — The standard error of the mean is actually the geometric standard error. (Observed vs Predicted)

4. Primary Outcome: Comparison of Observed and Predicted Trough Dabigatran Plasma Concentrations (C Trough,ss) at End of Trial (EoT) at Week 12
Description: Comparisons between dabigatran trough plasma levels as predicted by simulations to those observed in the study are performed to validate the dosing algorithm for Dabigatran Etexilate (DE).
  (As the trial was stopped prematurely, EOT may not be 12 weeks after randomisation for most of the patients)
  Despite the primary endpoint only being assessed in patients who received dabigatran etexilate, Warfarin was included as a comparator treatment in this study in order to facilitate informal comparisons of outcome events, and to look for efficacy signals in this previously unexplored population.
Time Frame: Week 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Observed | Predicted
Number analyzed (Participants) | 54 | 54
ng/mL | 108.21 (59.8) | 104.80 (59.8)
Statistical Analysis 1: Comparison: Observed vs Predicted; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; The Ctrough,ss (predicted or observed) was log transformed (natural logarithm) prior to fitting the ANOVA model; Adjusted Geometric Mean ratio = 103.25, 95% CI [86.40 to 123.40], Standard Error of Mean 1.11 — The standard error of the mean is actually the geometric standard error. (Observed vs Predicted)

5. Secondary Outcome: Percentage of Patients With Observed Trough Dabigatran Plasma Concentrations < 50 ng/mL at Week 1
Description: Percentage of patients with observed Ctrough,ss value < 50 ng/mL are presented. This outcome measure was only analysed for all patients together and not by dose group.
Time Frame: Week 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Patients Evaluated: All patients treated orally with either 150mg, 220mg or 300mg of dabigatran etexilate (DE) twice daily.
Arm/Group | Patients Evaluated
Number analyzed (Participants) | 130
percentage of participants | 26.9
Statistical Analysis 1: Comparison: Patients Evaluated; Test type: Superiority or Other; p < 0.001, Beta Function — Probability that P remains < 10% are presented, where P=Percentage of patients with observed Ctrough,ss value < 50 ng/mL; Probability calculated using Beta function ~B(1 + r, 1 + n - r),r=no. of patients(observed Ctrough,ss value < 50 ng/mL), n=no. of patients evaluated

6. Secondary Outcome: Percentage of Patients With Observed Trough Dabigatran Plasma Concentrations < 50 ng/mL at Week 2
Description: as for outcome 5
Time Frame: Week 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Patients Evaluated
Number analyzed (Participants) | 26
percentage of participants | 19.2
Statistical Analysis 1: Comparison: Patients Evaluated; Test type: Superiority or Other; p = 0.05, Beta Function — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]

7. Secondary Outcome: Percentage of Patients With Observed Trough Dabigatran Plasma Concentrations < 50 ng/mL at Week 4
Description: as for outcome 5
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Patients Evaluated
Number analyzed (Participants) | 112
percentage of participants | 9.8
Statistical Analysis 1: Comparison: Patients Evaluated; Test type: Superiority or Other; p = 0.46, Beta Function — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]

8. Secondary Outcome: Percentage of Patients With Observed Trough Dabigatran Plasma Concentrations < 50 ng/mL at End of Trial (EoT) Week 12
Description: Percentage of patients with observed Ctrough,ss value < 50 ng/mL (As the trial was stopped prematurely, EOT may not be 12 weeks after randomisation for most of the patients) This outcome measure was only analysed for all patients together and not by dose group.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Patients Evaluated
Number analyzed (Participants) | 54
percentage of participants | 7.4
Statistical Analysis 1: Comparison: Patients Evaluated; Test type: Superiority or Other; p = 0.65, Beta Function — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: From first intake of study drug until last intake of study drug plus 6 days (Up to 101 days).
Description: There were 8 patients who switched from dabigatran etexilate to warfarin during the study, and hence these patients are counted in the denominator of both arms. Any AEs which occurred in these patients are only presented under the treatment that the patient was taking at the time of the event.
Groups:
- Dabigatran Etexilate: Oral administration of 1 capsule of 150 mg (150 mg), 2 capsules of 110 mg (220 mg), or 2 capsules of 150 mg (300 mg) twice daily
Arm/Group | Dabigatran Etexilate | Warfarin
Serious Adverse Events (participants affected / at risk) | 19/162 | 11/89
Other Adverse Events (participants affected / at risk) | 64/162 | 38/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (N=162) | Warfarin (N=89)
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 1
Pericardial effusion (Cardiac disorders) | 5 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Device malfunction (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (N=162) | Warfarin (N=89)
Urinary tract infection (Infections and infestations) | 5 | 5
Dizziness (Nervous system disorders) | 3 | 5
Atrial fibrillation (Cardiac disorders) | 11 | 9
Pericardial effusion (Cardiac disorders) | 8 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Diarrhoea (Gastrointestinal disorders) | 19 | 2
Dyspepsia (Gastrointestinal disorders) | 15 | 0
Constipation (Gastrointestinal disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 5 | 5
Oedema peripheral (General disorders) | 10 | 2

LIMITATIONS AND CAVEATS:
This study was terminated prematurely due to safety concerns arising during conduct of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.